CLINICAL TRIAL: NCT05257031
Title: An Open-label, Non-Comparative, Multicentre Trial to Assess the Efficacy and Safety of SmofKabiven Extra Nitrogen for Parenteral Nutrition in Patients Receiving Intensive Care
Brief Title: Efficacy and Safety of SmofKabiven Extra Nitrogen for Parenteral Nutrition in Patients Receiving Intensive Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SKNt-002-CP3
Record Dates: First submitted 2022-01-31; First posted 2022-02-25 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Nutrition Therapy; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SmofKabiven extra Nitrogen (Experimental): The investigational product will be administered in a volume that provides the target caloric intake of 15 kcal/kg BW on Study Day 1 and 20 kcal/kg BW/day on Study Days 2 to 5.
  If calories are provided from other sources (e.g., enteral/oral nutrition/oral nutritional supplements or non-nutritional sources including glucose solution for drug dilution or propofol), the dose of the investigational product will be reduced accordingly to avoid calorie overload above the respective daily caloric targets.
  Interventions: Drug: SmofKabiven extra Nitrogen

INTERVENTIONS:
Drug: SmofKabiven extra Nitrogen — SmofKabiven extra Nitrogen contains amino acids (Aminoven®), glucose, lipids (SMOFlipid®: 30% soybean oil, 30% medium-chain triglycerides, 25% olive oil, 15% fish oil), and electrolytes.

SUMMARY:
The aim of this clinical trial is to assess the efficacy and safety of the investigational product SmofKabiven extra Nitrogen in patients requiring parenteral nutrition (PN) to achieve the target protein dose. The cumulative target protein dose is 6.2 g per kg of body weight (BW) over the five study treatment days, with 1.0 g/kg BW on Study Day 1 and 1.3 g/kg BW per day on Study Days 2-5; the target caloric intake is 15 kcal/kg BW on Study Day 1 and 20 kcal/kg BW/day on Study Days 2-5, following the recommendation of the ESPEN guideline on clinical nutrition in the intensive care unit 2019 regarding a slow-ramp up of calories during the first week of critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 90 years, male or female
* Critically ill, medical or surgical intensive care unit (ICU) patient
* The patient was admitted to the ICU during the previous 24-48 hours and has a minimum expected ICU stay of 5 days after the completion of screening
* Central venous access available for continuous infusion of the investigational product
* Contraindication against EN or limited tolerance to EN; it is planned that the patient receives ≥75% of the total target caloric intake from PN during the 5 investigational product treatment days
* Informed consent (signed and dated) from the patient to participate in this clinical trial. If the patient is unable to make a decision because of his/her critical condition, a decision regarding study enrolment is made at a case conference involving three physicians

Exclusion Criteria:

* Contraindication against PN or inability to receive PN via central venous access
* The patient has received PN within the last 7 days before the start of screening
* Body mass index (BMI) <18.5 kg/m2 or >35 kg/m2
* Any severe, persistent blood coagulation disorder with uncontrolled bleeding
* Any congenital errors of amino acid metabolism
* Uncontrolled hyperglycaemia despite insulin treatment
* Known hypersensitivity to fish, egg, soybean proteins, peanut proteins, or to any of the active ingredients or excipients contained in SmofKabiven extra Nitrogen
* General contraindications to infusion therapy: acute pulmonary oedema, hyperhydration, and decompensated cardiac insufficiency
* Severe renal insufficiency defined by the following criteria:

  * serum creatinine level > 353.6 µmol/L, or
  * creatinine level ≥ 3.0 times higher than the upper limit of normal (according to the KDIGO 2012 Clinical Practice Guideline), or
  * diuresis < 0.3 mL/kg/hr during ≥ 12 hrs (Acute Kidney Injury stage ≥ 3 according to the KDIGO 2012 Clinical Practice Guideline) without access to renal replacement therapy
* Unstable haemodynamic conditions (e.g., acute myocardial infarction, stroke, embolism, severe sepsis, shock) including acute shock (arterial serum lactate > 2.0 mmol/L)
* Severe liver insufficiency
* Haemophagocytic syndrome
* Pregnancy or lactation
* Receiving end-of-life care
* Severe hyperlipidaemia (serum cholesterol and/or triglycerides and/or LDL-C level at least 1.5 times higher than the upper limit of normal range)
* Pathologically elevated serum levels of any of the included electrolytes (sodium, potassium, magnesium, total calcium, chloride, inorganic phosphate)
* Participation in another interventional clinical trial within the previous 4 weeks
* Previous inclusion in the present study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Protein intake during the study treatment period | Study Days 1 to 5
  Percentage of patients who have reached ≥ 70% of the cumulative target protein intake.

SECONDARY OUTCOMES:
Percentage of the cumulative target protein intake reached over the study treatment period | Study Days 1 to 5
Mean daily protein intake from parenteral nutrition (PN), enteral nutrition (EN), oral nutrition (ON), oral nutrition supplements (ONS) over the study treatment period | Study Days 1 to 5
Cumulative protein intake from PN, EN, ON, ONS over the study treatment period | Study Days 1 to 5
Mean daily caloric intake from PN, EN, ON, ONS, and non-nutritional sources over the study treatment period | Study Days 1 to 5
Cumulative caloric intake from PN, EN, ON, ONS, and non-nutritional sources over the study treatment period | Study Days 1 to 5

OTHER OUTCOMES:
Incidence of adverse events | Until 24 hours after the end of last infusion
Incidence of serious adverse events | Until 24 hours after the end of last infusion
Changes in vital signs (blood pressure) | Study Days 1 to 6
Changes in vital signs (heart rate) | Study Days 1 to 6
Changes in vital signs (respiratory rate) | Study Days 1 to 6
Changes in vital signs (body temperature) | Study Days 1 to 6
Adverse events of special interest: hyperglycaemia, hypoglycaemia, hypertriglyceridemia | Until 24 hours after the end of last infusion
Changes in laboratory variables (number of patients with abnormal values) | Study Days 4 and 6
Incidence of (serious) adverse events | 24 hours after the end of the last infusion up to Study Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Denis N Protsenko, MD, Principal Investigator — Municipal Clinical Hospital No. 40 of Moscow Healthcare Department
Locations (1):
- Municipal Clinical Hospital No. 40 of Moscow Healthcare Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No